CLINICAL TRIAL: NCT06344533
Title: Phase I Clinical Study to Evaluate the Safety, Tolerability, and Pharmacokinetic Characteristics of JMKX003142 Injection Administered Randomly, Double-blind, Placebo-controlled, Single-ascending Dose and Multiple-ascending Doses in Chinese Healthy Adult Subjects
Brief Title: Study of JMKX003142 Injection in Chinese Healthy Subjects
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Jemincare (Industry)
Collaborators: Zhejiang Hangyu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: JMKX003142iv-101
Record Dates: First submitted 2024-03-18; First posted 2024-04-03 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-03

CONDITIONS: Healthy Adult

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- JMKX003142 Injection (Experimental): Single and multiple doses of JMKX003142 Injection administered intravenously.
  Interventions: Drug: JMKX003142 Injection
- Placebo (Placebo Comparator): Placebo administered intravenously.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: JMKX003142 Injection — JMKX003142 Injection will be administered intravenously once in SAD cohorts and once daily in MAD cohorts for 5 consecutive days.
  Arms: JMKX003142 Injection
Drug: Placebo — Matching placebo will be administered intravenously once in SAD cohorts and once daily in MAD cohorts for 5 consecutive days.
  Arms: Placebo

SUMMARY:
To Evaluate the Safety, Tolerability, and Pharmacokinetic Characteristics of JMKX003142 Injection Administered Randomly, Double-blind, Placebo-controlled, Single-ascending Dose and Multiple-ascending Doses in Chinese Healthy Adult Subjects

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects aged 18-45 years (including boundary values).
2. Able to sign a written informed consent form.
3. Physical examination, clinical laboratory examination value, Virology examination, vital signs and ECG examination are confirmed by the researcher to be normal or abnormal without clinical significance
4. The subjects have a thorough understanding of the study content, process, and potential adverse effects, and are willing to complete the study according to the requirements of the experimental protocol

Exclusion Criteria:

1. Had or currently have serious clinical diseases related to circulatory system, respiratory system, digestive system, nervous system, endocrine system, blood lymphatic system, genitourinary system or psychiatry, as well as habitual constipation, gastrointestinal bleeding history, which is judged to be inappropriate for the study by the investigators
2. Participants in any other clinical study within 3 months prior to the first administration of this study
3. The investigators believe that the subject has other factors that are not suitable for participating in this experiment
4. Pregnant or lactating women

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 78 (Estimated)
Dates: Start 2024-04-10 (Estimated); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
Number of the Adverse Events that are related to the single dose treatment | From Baseline to Day7
  single dose safety single dose safety
Number of the Adverse Events that are related to the multiple dose treatment | From Baseline to Day12
  multiple dose safety multiple dose safety

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No